CLINICAL TRIAL: NCT06826703
Title: the Effect of Motivational Interviewing Based on Health Promotion Model on Diabetes Self-management and Cyberchondria Severity in Individuals With Diabetes
Brief Title: The Effect of Motivational Interviewing on Diabetes Self-Management and Severity of Cyberchondria in Individuals With Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Gülşen Altuntas Çalım, health services teacher in the ministry of national education, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AU-SBF-GAÇ-02
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes; Motivation; Self-management
Keywords: cyberchondria violence; health belief model; self-management; type 2 diabetes; motivational interview
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: the experimental group will be trained with motivational technique. the control group will not receive any intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group receiving diabetes education with motivational interviewing technique based on health belief m (Experimental): Patient Introduction Form, Diabetes Self-Management Scale (DSMS), Cyberchondria Severity Scale-Short Form (CSS-SS-SF) scales will be applied to the experimental group before the training. Then, individuals in the experimental group will be given diabetes education one day a week with the motivational interviewing technique based on the health belief model. A total of 4 weeks of education will be given. After the end of the training, Patient Introduction Form, Diabetes Self-Management Scale (DMSS), Cyberchondria Severity Scale-Short Form (SCS-SF) scales will be applied.
  Interventions: Other: Experimental Group
- group who did not receive diabetes education with motivational interviewing technique (No Intervention): Patient introduction form, Diabetes Self-Management Scale (DMSMS), Cyberchondria Severity Scale-Short Form (CSS-SS-SF) scales will be applied to the control group at the first encounter. After 1 month, the Patient Introduction Form, Diabetes Self-Management Scale (DMSS), Cyberchondria Severity Scale-Short Form (CSS-SF) scales will be applied again. No application will be made to the control group

INTERVENTIONS:
Other: Experimental Group — Individuals will receive diabetes education with motivational interviewing technique based on health belief model.
  Arms: group receiving diabetes education with motivational interviewing technique based on health belief m

SUMMARY:
Objective: The aim of this study was to determine the effects of diabetes education given to individuals with diabetes using motivational interviewing technique based on the health promotion model on diabetes self-management and cyberchondria severity. Materials and Method: The population of the study consisted of 1000 individuals. The sample consisted of 64 individuals, 32 experimental and 32 control, who met the research criteria. The research will be conducted between 15.02.2025-15.03.2025 in Van Regional Training and Research Hospital Diabetes outpatient clinic. Data in the research; Descriptive Information Form, Diabetes Self-Management Scale (DMS), Cyberchondria Severity Scale-Short Form (CSS-SF) scales will be applied. Research experiment Motivational interviewing intervention based on the health belief model will be conducted once a week for 1 month. At the end of 1 month, both scales will be administered again to individuals in both experimental and control groups.

DETAILED DESCRIPTION:
Objective: The aim of this study is to determine the effects of diabetes education given to individuals with diabetes using motivational interviewing technique based on the health promotion model on diabetes self-management and cyberchondria severity. Material and Method: The population of the study consisted of 1000 individuals. The sample consisted of 64 individuals, 32 experimental and 32 control, who met the research criteria. The research will be conducted in Van Regional Training and Research Hospital Diabetes outpatient clinic between 15.02.2025-15.03.2025. Data in the study; Descriptive Information Form, Diabetes Self-Management Scale (DMSS), Cyberchondria Severity Scale-Short Form (CSS-SF) scales will be applied. Research experiment The motivational interviewing intervention based on the health belief model will be conducted once a week for 1 month. At the end of 1 month, both The scales will be administered again to the individuals in both the experimental group and the control group. Descriptive statistical methods (number, percentage), chi-square test, independent t-test in groups and paired t-test will be used.

ELIGIBILITY:
Inclusion Criteria:

* Having diabetes for at least 6 months
* Being over 18 years old
* To have sufficient communication skills to answer verbal and written questions and fulfill instructions
* Being literate
* No physical, cognitive or mental impairment in answering the questions
* Willingness to participate in research.

Exclusion Criteria:

* Being under 18 years of age
* Being hospitalized in inpatient treatment institutions due to DM or DM complications during the research process
* The emergence of any health problem that prevents the person from continuing the research
* Do not leave the study voluntarily.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Cyberchondria Severity Scale-Short Form (CSS-SF) | one months
  The scale assesses the severity of cybercronyism. Items can be summed to form a total score. The lowest score that can be obtained from the scale is 0 and the highest score is 60.It consists of 12 items.
  * Extremism The incremental and repetitive nature of research 1, 3, 6
  * Anxiety Anxiety/anxiety as a result of research 4, 8, 9
  * Assurance Research that encourages individuals to seek professional medical advice 5, 11, 12
  * Coercion Web searches affecting all aspects of life 2, 7, 10
Diabetes Self-Management Perception Scale (DSMAS) | one month
  The scale consists of 8 items. PERCEPTION OF SELF-MANAGEMENT IN DIABETES SCALE (DÖYAS)
  Choose the option closest to you... Strongly disagree............. . (1) Disagree with ........................ ... (2) Undecided................................ (3) Agree......................... .... (4) Strongly agree...................(5) The minimum score that can be obtained from the scale is 8 and the maximum score is 40.. A high total score indicates that the individual's awareness in diabetes management is very good

CONTACTS AND LOCATIONS:
Locations (1):
- Van Regional Training and Research Hospital Diabetes Polyclinic, Van, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No